CLINICAL TRIAL: NCT02927899
Title: Acceptability in the Taste of Tomato-Soy-Arugula Seed Beverages in Men With Prostate Cancer
Brief Title: Taste Acceptability of Tomato-Soy-Arugula Seed Beverages in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-15064; NCI-2016-01252 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Prostate Carcinoma
Keywords: Tomato-Soy-Arugula
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (dietary intervention, survey) (Experimental): Patients receive 4 tomato-soy beverages and 3 labeled arugula seed powder portions. Patients add 1 arugula seed powder portion to each of 3 tomato-soy beverages immediately prior to consumption, and they consume 1 beverage without the powder. After each beverage tasting, patients complete a survey on the sensory acceptability of the sample.
  Interventions: Other: Survey Administration; Dietary Supplement: Tomato-Soy Juice

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Dietary Supplement: Tomato-Soy Juice — Receive tomato-soy beverages with or without varying levels of arugula seed powder

SUMMARY:
This study is a sensory analysis of several different formulations of a novel tomato-soy-arugula seed beverage in men with prostate cancer. Eating a diet rich in a variety of fruits and vegetables has been associated with decreased risk of a variety of diseases, including prostate cancer. Mixed vegetable beverages may be useful in prostate cancer survivorship.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the sensory acceptability of a novel tomato-soy-arugula seed beverage in men with prostate cancer.

OUTLINE:

Patients receive 4 tomato-soy beverages and 3 labeled arugula seed powder portions. Patients add 1 arugula seed powder portion to each of 3 tomato-soy beverages immediately prior to consumption and they consume 1 beverage without the powder. After each beverage tasting, patients complete a survey on the sensory acceptability of the sample.

ELIGIBILITY:
Inclusion Criteria:

* Have a prostate cancer diagnosis
* Not be allergic to tomato or tomato products
* Not be allergic to soy or soy related products
* Not be allergic to any cruciferous vegetables (e.g.: broccoli, cauliflower, kale, brussels sprouts, arugula/rocket, bok choy, etc.)
* Voluntarily agree to participate and read the informed consent documents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
Sensory acceptability of tomato-soy-arugula seed beverages assessed by survey | Up to 2 years
  Mean plus/minus standard deviation will be used to express the results from the acceptability tests and the Just About Right tests. Ranking results will be analyzed by using t-test to obtain determine statistical significance. Significance level of the value will be chosen before statistic tests are conducted, at a value of 5%. A critical value below p < 0.05, will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu